CLINICAL TRIAL: NCT05838807
Title: The Effects of Thermal and Pulsed Ultrasound on Pain and Function in Individuals With Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Thermal and Pulsed Ultrasound for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/004245
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome; Median Neuropathy, Carpal Tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: The study will be a level II randomized controlled trial with a parallel group design. Participants will be randomized to receive one of four interventions: thermal ultrasound, pulsed ultrasound, a combination of both, or a placebo treatment. Participants will receive their assigned treatment for 10 minutes, three times per week, for 4 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to the participants being blinded to the treatment they are receiving, the outcome assessors will also be blinded to the treatment assignment. This will ensure that the assessors are unbiased when measuring the outcome measures of pain intensity, functional status, and nerve conduction studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Thermal Ultrasound Group (Experimental)
  Interventions: Device: Thermal Ultrasound
- Group B: Pulsed Ultrasound Group: (Experimental)
  Interventions: Device: Pulsed Ultrasound
- Group C: Combination Group (Experimental)
  Interventions: Device: Combined Ultrasound
- Group D: Placebo Group (Placebo Comparator)
  Interventions: Device: Placebo Ultrasound

INTERVENTIONS:
Device: Thermal Ultrasound — Participants in this group will receive thermal ultrasound treatment using a gel-coupled ultrasound probe that delivers continuous ultrasound waves at a frequency of 1 Mega Hertz. The ultrasound probe will be moved continuously over the affected wrist and hand region for 5 minutes per session, three times per week, for four weeks. The intensity of the ultrasound wave will be set at 1.0 W/cm2 applied for 5 minutes. The treatment will be administered three times per week, for four weeks.
  Arms: Group A: Thermal Ultrasound Group
Device: Pulsed Ultrasound — Participants in this group will receive pulsed ultrasound treatment using a gel-coupled ultrasound probe that delivers pulsed ultrasound waves at a frequency of 1 Mega Hertz. The ultrasound probe will be moved continuously over the affected wrist and hand region for 15 minutes with 25% duty cycle and intensity of 1.0 W/cm2.The treatment will be administered three times per week, for four weeks.
  Arms: Group B: Pulsed Ultrasound Group:
Device: Combined Ultrasound — Participants in this group will receive a combination of thermal and pulsed ultrasound treatments. The thermal ultrasound treatment will be administered first for 5 minutes, followed by the pulsed ultrasound treatment for another 15 minutes. The same parameters as described above will be used for each treatment modality. The combination treatment will be administered three times per week, for four weeks.
  Arms: Group C: Combination Group
Device: Placebo Ultrasound — Participants in this group will receive a placebo ultrasound treatment that looks and feels identical to the active ultrasound treatments, but does not deliver any therapeutic effects. The placebo treatment will be administered using the same gel-coupled ultrasound probe for 15 minutes per session, three times per week, for four weeks, with the intensity set at 0 W/cm² and the temperature maintained at room temperature.
  Arms: Group D: Placebo Group

SUMMARY:
This study will be a Randomized controlled trial with a sample size of at least 100 individuals with carpal tunnel syndrome. Participants will be randomized to receive either thermal ultrasound, pulsed ultrasound, a combination of both, or a placebo treatment for 10 minutes, three times per week, for 4 weeks. Outcome measures will include pain intensity, functional status, and nerve conduction studies. Outcome measures will be assessed at baseline, 4 weeks, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 30-60 years old
2. Diagnosis of carpal tunnel syndrome based on clinical symptoms and nerve conduction studies, including:

   * Symptoms of pain, numbness, and tingling in the hand and/or fingers, particularly the thumb, index, and middle fingers
   * Positive Tinel's sign (tapping over the median nerve at the wrist elicits tingling or numbness in the hand)
   * Positive Phalen's maneuver (flexion of the wrist for 60 seconds elicits tingling or numbness in the hand)
   * Abnormal nerve conduction studies showing prolonged distal motor latency, and/or decreased amplitude of the median nerve

Exclusion Criteria:

1. Prior surgery for carpal tunnel syndrome
2. History of wrist or hand fracture in the past year
3. Pregnancy or planning to become pregnant during the study period
4. Active infection or skin condition in the treatment area
5. Known allergy to ultrasound gel or other components of the treatment
6. Use of corticosteroids or other medications that may affect nerve function within the past 3 months
7. Participation in another clinical trial within the past 30 days

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Changes in pain intensity at baseline, 4 weeks after randomization, and 8 weeks after discharge.
  This will be measured using the visual analogue scale (VAS), which is a valid and reliable tool for assessing pain intensity. The VAS is a 10-cm horizontal line with anchors of "no pain" and "worst pain imaginable," and participants will be asked to mark their level of pain intensity on the line.
Functional Status | Changes in functional status at baseline, 4 weeks after randomization, and 8 weeks after discharge.
  his will be measured using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, which is a validated instrument for assessing upper extremity function. The DASH consists of 30 items assessing physical function, symptoms, and social-emotional aspects of disability, and scores range from 0 (no disability) to 100 (severe disability).

SECONDARY OUTCOMES:
Nerve Conduction Studies | Changes in nerve conduction studies at baseline, 4 weeks after randomization, and 8 weeks after discharge.
  This will be assessed using nerve conduction studies (NCS), which are a validated tool for assessing nerve function in individuals with carpal tunnel syndrome. NCS will be used to measure median nerve sensory and motor distal latency in addition to the amplitude of the median nerve.
Hand grip strength | Changes in hand grip strength at baseline, 4 weeks after randomization, and 8 weeks after discharge.
  This will be measured using a handheld dynamometer, which is a validated tool for assessing grip strength in individuals with carpal tunnel syndrome. Participants will be asked to squeeze the dynamometer as hard as possible, and the highest value of three trials for each hand will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be available upon reasonable request. Requests for access to the data should be submitted via email to mohamed.elmeligie@acu.edu.eg. All requests will be reviewed by the study investigators to ensure that they are reasonable and consistent with the ethical principles of the study. Access to the data will be granted in compliance with applicable laws and regulations, and with appropriate safeguards to protect the privacy and confidentiality of study participants.
Supporting Information: SAP, ICF
Time Frame: During the trial and 1 year after the trial end.
Access Criteria: via email to mohamed.elmeligie@acu.edu.eg

REFERENCES:
- [Derived] ElMeligie MM, Ismail MM, Yehia AM, Sakr HR, Amin DI. Effects of Thermal and Pulsed Ultrasound on Pain and Function in Patients With Carpal Tunnel Syndrome: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Jun 1;104(6):e83-e91. doi: 10.1097/PHM.0000000000002651. Epub 2024 Nov 11. PMID 39773605